CLINICAL TRIAL: NCT02939846
Title: A Phase I Study to Evaluate the Pharmacokinetics and Safety of Single and Repeat Oral Doses of Trametinib in Chinese Subjects With Solid Tumours
Brief Title: Pharmacokinetics of Single and Repeat Oral Doses of Trametinib in Chinese Subjects With Solid Tumours
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in strategy
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201021
Record Dates: First submitted 2015-05-07; First posted 2016-10-20 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2017-01

CONDITIONS: Cancer
Keywords: Safety; Solid tumor; Trametinib; Pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trametinib (Experimental): Subjects will be administrated with trametinib 2 mg once daily until disease progression.
  Interventions: Drug: Trametinib

INTERVENTIONS:
Drug: Trametinib — Trametinib study will be provided as 0.5 mg and 2.0 mg tablets. Each tablet will contain 0.5 mg or 2.0 mg of trametinib parent (present as the DMSO solvate)

SUMMARY:
Present clinical study will be conducted in China to evaluate the pharmacokinetics of single and repeat oral doses of trametinib, the safety profile and the clinical activity in Chinese subjects with solid tumor. Approximately 10 evaluable subjects will be enrolled in the study, Subjects will receive trametinib 2 mg once daily (QD). Study treatment will continue until disease progression, death or unacceptable toxicity. The study will be completed after all subjects have discontinued from study treatment or last enrolled subject has had at least 16 weeks of follow-up, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed written informed consent
* Males and females ≥18 years of age (at the time consent is obtained).
* Histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumours, melanoma subjects will be eligible if BRAF V600 mutation was confirmed in the tumour tissue by qualified clinical laboratories. The disease is not responsive to standard therapies, or for which there is no approved or curative therapy.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Adequate baseline organ function defined by: Absolute neutrophil count (ANC): >=1,200 /microliter (uL); Hemoglobin: >=9 grams (g)/deciliter (dL); Platelets: >=75,000 /uL; Prothrombin time/ International normalization ratio and activated partial thromboplastin time: <=1.5 x Upper Limit of Normal (ULN); Total bilirubin: <=1.5 x ULN; Aspartate aminotransferase and Alanine aminotransferase: <=2.5 x ULN; Calculated creatinine clearance (Calculate creatinine clearance using standard Cockcroft-Gault formula): >=50 milliliter (mL)/ minute (min) or 24-hour urine creatinine clearance>=50 mL/min; Left ventricular Ejection fraction (LVEF): >/= 50% LVEF in case there is no established Lower limit of normal (LLN) for a given institution.
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels. Subjects with prior Whipple procedure (pancreaticoduodenectomy) are eligible (if meeting above criteria).
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from the time of the first dose of trametinib until 16 weeks after the last dose of trametinib.
* Women of child-bearing potential must have a negative serum pregnancy test within 7 days of first dose of study treatment and agree to use effective contraception from 14 days prior to enrolment, throughout the treatment period and for 4 months after the last dose of study treatment.

Exclusion Criteria:

* Pregnant or Lactating female.
* History of another malignancy. Exception: Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Use of an investigational drug within 28 days or five half-lives, whichever is longer preceding the first dose of trametinib.
* Previous treatment with a MEK inhibitor.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or sub-investigator, contraindicates their participation.
* History of interstitial lung disease or pneumonitis.
* Current use of a prohibited medication as described in Section 10.2.

  •Colony-stimulating factors like filgrastim are prohibited during treatment as a prophylactic management.
* Any major surgery, radiotherapy, or immunotherapy within 21 days before initiation of trametinib. Chemotherapy regimens with delayed toxicity within 21 days before initiation of trametinib (42 days for prior nitrosourea or mitomycin C). Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the two weeks before initiation of trametinib.

Note: Use of bisphosphonates is considered supportive care and their use is permitted.

* History or current evidence / risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR):

  * Uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes).
  * Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or CSR such as:
  * Evidence of new optic disc cupping
  * Evidence of new visual field defects on automated perimetry
  * Intraocular pressure > 21mm Hg as measured by tonography
* Symptomatic or uncontrolled leptomeningeal or brain metastases or spinal cord compression.

  * Subjects previously treated for these conditions that have had stable central nervous system (CNS) disease are asymptomatic and off corticosteroids, or are on stable dose of corticosteroids for at least 1 month prior to study Day 1 are eligible.
  * Subjects are not eligible to receive enzyme inducing anti-epileptic drugs (EIAEDs).
* QTc B ≥ 480 msecs.
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks.
* History or evidence of current ≥ Class II congestive heart failure as defined by New York Heart Association.
* History or evidence of current clinically significant uncontrolled arrhythmias.

  • Subjects with controlled atrial fibrillation for >1 month prior to study Day 1 are eligible.
* History of Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection.

  • Subjects with laboratory evidence of cleared HBV and/or HCV will be permitted, which defined as HBs antigen negative and HBV DNA negative(HBV DNA result is mandatory if both or either HBc and HBs antibody is positive); and HCV antibody is negative.
* History of HIV infection.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease).
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to dimethyl sulfoxide (DMSO).
* Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
PK parameters of trametinib following single and repeat dose(2mg QD): Cmax | At Day 1:Pre-dose, 0.5hr,1hr, 2hr,3hr,4hr, 6hr,10hr,24hr
PK parameters of trametinib following single and repeat dose(2mg QD): Tmax | At Day 1:Pre-dose, 0.5hr,1hr, 2hr,3hr,4hr, 6hr,10hr,24hr
PK parameters of trametinib following single and repeat dose(2mg QD): AUC (0-24h) | At Day 1:Pre-dose, 0.5hr,1hr, 2hr,3hr,4hr, 6hr,10hr,24hr
PK parameters of trametinib following single and repeat dose(2mg QD): Cmin.ss | At Day 22:Pre-dose, 0.5hr,1hr, 2hr,3hr,4hr, 6hr,10hr,24hr
PK parameters of trametinib following single and repeat dose(2mg QD): Cmax.ss | At Day 22:Pre-dose, 0.5hr,1hr, 2hr,3hr,4hr, 6hr,10hr,24hr
PK parameters of trametinib following single and repeat dose(2mg QD): Cavg.ss | At Day 22:Pre-dose, 0.5hr,1hr, 2hr,3hr,4hr, 6hr,10hr,24hr
PK parameters of trametinib following single and repeat dose(2mg QD): AUC(0-24h) | At Day 22:Pre-dose, 0.5hr,1hr, 2hr,3hr,4hr, 6hr,10hr,24hr
Accumulation ratio of trametinib following single and repeat dose(2mg QD) | At Day 22
Effective half-life of trametinib following single and repeat dose(2mg QD) | At Day 22

SECONDARY OUTCOMES:
Composite of Physical examination assessment | Up to 30 days of the subject's last dose
  Physical examination will include assessments of eyes, neurological and cardiovascular systems, lungs, abdomen, head, neck, ears, nose, mouth, throat, thyroid, lymph nodes, extremities, and skin, genitourinary (pelvic) and rectal exams.
Composite of Safety and tolerability as assessed by vital signs assessment: blood pressure, temperature and pulse rate | Up to 30 days of the subject's last dose.
  Vital sign measurements will include systolic and diastolic blood pressure, body temperature and pulse rate.
Electrocardiogram (ECG) assessment | Every week in the 1st month, week 8, and then every 8 weeks until treatment discontinuation up to 30 days of the subject's last dose (assessed up to 5 years)
  12-lead ECGs will be obtained at each time point using an ECG machine that automatically to calculate the heart rate and measures PR, QRS, QT and corrected QT interval duration (QTc intervals).
Echocardiogram (ECHO) assessment | At week 4, week 8, and then every 8 weeks until treatment discontinuation up to 5 years
  ECHO assessment will include an evaluation for left ventricular ejection fraction.
Eye exams assessment | At screening, and when clinical indicated until treatment discontinuation up to 5 years
Chemistry laboratory values assessment | Up to 30 days of the subject's last dose.
Number of subjects with Adverse events (AEs) | Up to 30 days of the subject's last dose.
Number of subjects with Serious Adverse events (SAEs) | Up to 30 days of the subject's last dose.
Objective response rate (ORR) | Every 2 months until disease progression up to 5 years
  ORR defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation
Progression free survival(PFS) | Every 2 months until disease progression up to 5 years
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause
Hematology laboratory values assessment | Up to 30 days of the subject's last dose
Urinalysis laboratory values assessment | Up to 30 days of the subject's last dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline